CLINICAL TRIAL: NCT05736588
Title: A Stigma Responsive Service Delivery Model for HPV-based Screening Among Women Living With HIV
Brief Title: Elimisha HPV (Human Papillomavirus)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00111929; 1R01TW012415 (NIH)
Record Dates: First submitted 2023-02-08; First posted 2023-02-21 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Cervical Cancer; HPV; HIV; Stigma
MeSH Terms: conditions — Uterine Cervical Neoplasms; Social Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention)
- Elimisha HPV (Experimental): Elimisha HPV is a multi-level stigma-responsive cervical cancer prevention service delivery model that incorporates stigma-responsive education, peer navigation and a patient-centered delivery strategy, addressing drivers while mitigating harms from stigma.
  Interventions: Behavioral: Elimisha HPV

INTERVENTIONS:
Behavioral: Elimisha HPV — Elimisha HPV is a multi-level stigma-responsive cervical cancer prevention service delivery model that incorporates stigma-responsive education, peer navigation and a patient-centered delivery strategy, addressing drivers while mitigating harms from stigma.
  Arms: Elimisha HPV

SUMMARY:
This research study aims to develop a stigma-responsive educational intervention which includes simplified scripts that provide clear messages about HPV and video aimed at addressing fears and misperceptions from a peer perspective. These educational components will be incorporated into 'Elimisha' HPV a multi-level stigma-responsive cervical cancer prevention service delivery model.

DETAILED DESCRIPTION:
4.1.a. Detailed Description To determine the impact of this intervention on cervical cancer screening uptake and treatment we will carry out a cluster-RCT in community health units (CUs) nested within 12 government-supported health facilities. Over a twelve-month period, Community Health Volunteers within the CUs will offer HPV-based cervical cancer screening during routine home visits, coupled with themocoagulation free-of-charge by the providers in the parent health facility. Screening will be offered using the current standard of care model or using the enhanced Elimisha intervention, according to their assigned arm, described below.

Control: CUs in control areas will offer HPV-testing via self-collection to all women in their catchment population using a standard of care model. Screening activities will be carried out by ten CHVs per facility, comprising one CU. CHVs within each CU will be overseen by their CU supervisor. CHVs will lead outreach and education activities, and individual counseling about HPV-testing during routine home visits, including instructions about self-collection, and processing of the specimens. Within two weeks, laboratory results will be sent to the CHVs to record in the facility register and notify women via text, phone call or home visit. Women who test positive for HPV will be referred to their parent health facility for visual inspection with acetic acid, followed by treatment with thermocoagulation as indicated, the current standard of care. Women with lesions not amenable to treatment with thermocoagulation will undergo loop electrosurgical excision procedure at the same visit. Women with lesions suspicious for cancer will undergo biopsy and have follow-up with the gynecologist at the district hospital for treatment planning. Women who are delayed in seeking follow-up (greater than three months since notification of diagnosis) will receive additional text message reminders and home visits, per clinic protocol.

Elimisha HPV: a multi-level stigma-responsive delivery model for HPV-based cervical cancer screening (intervention): CHVs in community health units in the intervention arm will offer HPV-testing along with the additional components of Elimisha HPV. CHVs who have been trained in patient-centered care will provide education using standardized scripts reviewed to ensure content is not stigmatizing. For women not ready to screen at this point, counseling will be followed by a brief educational video in which a peer describes her experience with screening and treatment. Will will be provided an illustration to describe the self-sampling procedure. Laboratory process time and notification of results is the same as in control facilities. Women who decline screening will be offered the option to be linked with a peer supporter, who will reach out to her within the following week. Women who are delayed in seeking follow-up care will receive a phone call from a peer support person, who will offer to discuss how own experience and answer any questions about treatment process.

Follow-up administration of stigma measurement tool: In months 9-12 of the c-RCT, the study team will recruit women attending study health facilities in both arms to complete the validated instrument to measure HPV, HIV and cervical cancer-related stigma. We will randomly select women who have completed their routine visits with the assumption that after that point in the study, they will have had exposure to the assigned cervical cancer screening delivery strategy, and for those who have tested positive for HPV, will have had time to follow-up for treatment. Women will be considered eligible if they are in the age eligibility range for cervical cancer screening (30-65), but may or may not report that they have been offered or accepted screening as that will be evaluated as an outcome. The instrument contains approximately 55 items, and will take 30 minutes to complete. Instruments have been translated and validated into Dhluo, and will be administered orally with computer-assisted answer entry to ensure confidentiality.

3618 women were screened for HPV but were not consented as the screening was part of their clinical care. 982 participants, including some women screened, and community health promoters (CHP) and CHP supervisors, consented to the study to complete the surveys and in depth interviews.

ELIGIBILITY:
Aim 2 Participants Women registered within the 12 community units participating in the study (Aim 2)

For Aim 2, activity 4, we will enroll approximately 804 randomly selected women, (67 per community unit in each of 12 facilities)

Inclusion criteria:

* A Community Health Volunteer (CHV) has registered the woman in the mSaada App (electronic HPV-based cervical cancer screening tracking tool) during the study period
* Is eligible for cervical cancer screening per the Kenya Ministry of Health guidelines include:

  * Women living with HIV (WLWH) will be between the age of 25 and 65
  * All other women will be between the age of 30 and 65
  * All women should have an intact uterus and cervix

Exclusion criteria:

* Does not understand the study purpose and details
* Is not willing to provide informed consent

CHVs working through government-supported health facilities (Aim 2) We will work with CHV supervisors to approach CHVs for study participation and possible enrollment into the study for training and participation in the stigma-responsive service delivery model. Since study outcomes may appear to reflect CHV job performance, we will explain this as part of the informed consent and emphasize the voluntary nature of participation in the study. For both optimization of study activities and to avoid any coercion, CHVs will be able to decline participation without impact on their position in the facility.

Inclusion criteria:

* Age 18 or older
* Must be a Community Health Volunteer (CHV) at government-supported facilities in Kisumu County

Exclusion criteria:

* Does not understand the study purpose and details
* Is not willing to sign an informed consent

Aim 3 Participants Participants will be purposively recruited from each study arm to achieve a sample with heterogeneous demographic and clinical characteristics (e.g., age, HIV and HPV status).

Women attending government-supported health facilities (Aim 3) Investigators will enroll approximately 24 women with the option to recruit more if new themes are emerging in the IDIs.

Inclusion criteria:

* Will have completed an HPV screening test at one of the intervention or control facilities
* Agree to be audio recorded

Exclusion criteria:

* Does not understand the study purpose and details
* Is not willing to provide informed consent

Community Health Volunteers (CHVs) and Peer Navigators (Aims 3) Investigators will enroll approximately 10 CHVs and peer navigators with the option to recruit more if new themes are emerging in the IDIs.

Inclusion criteria:

* Participated as a CHV or peer navigator at one of the facilities participating in the study
* Agree to be audio recorded

Exclusion criteria:

* Does not understand the study purpose and details
* Is not willing to sign an informed consent

Facility managers (Aim 3) Investigators will enroll approximately 12 facility managers.

Inclusion criteria:

* Age 18 or older
* A manager at one of the facilities participating in the study
* Agree to be audio recorded

Exclusion criteria

* Does not understand the study purpose and details
* Is not willing to sign an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 982 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2024-11-26 (Actual)

PRIMARY OUTCOMES:
Overall HPV testing rates | 1 day
  Number of women screened for HPV/Number of women eligible for HPV-based cervical cancer screening during study period

SECONDARY OUTCOMES:
HPV testing rates among women living with HIV (WLWH) enrolled in HIV care | 1 day
  Number of WLWH enrolled in HIV care screened for HPV/Number of WLWH living in the study area
Follow-up rates for HPV treatment | 1 day
  Number of women testing HPV+ seeking treatment within 3 months/Number of women testing HPV+
Follow-up rates for HPV treatment among WLWH | 1 day
  Number of WLWH testing HPV+ seeking HPV treatment within 3 months/Number of WLWH testing HPV+
Proportion of WLWH enrolled in HIV care attending at least one visit within study period | 1 day
  Proportion of WLWH enrolled in HIV care attending at least one visit within study period
Overall level of stigma related to cervical cancer, HPV and HIV | 1 day
  HPV and Cervical Cancer Associated Stigma Scale will be used which is scored on a scale of 0 (strongly disagree) to 3 (strongly agree) within each health domain.
Level of stigma related to cervical cancer | 1 day
  HPV and Cervical Cancer Associated Stigma Scale will be used which is scored on a scale of 0 (strongly disagree) to 3 (strongly agree) within cervical cancer domain
Level of stigma related to HPV | 1 day
  HPV and Cervical Cancer Associated Stigma Scale will be used which is scored on a scale 0 (strongly disagree) to 3 (strongly agree) within HPV domain.
Level of stigma related to HIV | 1 day
  HPV and Cervical Cancer Associated Stigma Scale will be used which is scored on a scale of 0 (strongly disagree) to 3 (strongly agree) within HIV domain.

OTHER OUTCOMES:
Factors related to the success of the delivery model | 1 day
  Factors at the patient, community health volunteer and peer navigator level; factors at the health facility level; and factors at the County Health Management Team level.

CONTACTS AND LOCATIONS:
Locations (1):
- Kenya Medical Research Institute, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF

DOCUMENTS (1):
  • Informed Consent Form (2024-03-28): https://cdn.clinicaltrials.gov/large-docs/88/NCT05736588/ICF_000.pdf